CLINICAL TRIAL: NCT06804291
Title: The Effect of Different Exercise Modes on Serum Concentrations of NfL, APP, and BLBP: a Nonrandomized Control Trial Exploratory Study
Brief Title: The Effect of Cycling, Running, and Playing Rugby on Three Biomarkers That May Indicate Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Principal Investigator, Matthew Rogatzki, Assistant Professor, Appalachian State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-0286
Record Dates: First submitted 2025-01-25; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Male and Female Subjects
Keywords: Brain injury biomarkers
MeSH Terms: interventions — Running; Jogging; albumin Rugby Park; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Running Group (Active Comparator): Participants run 6.44 kilometers. Venous blood is drawn prior to the run, immediately after the run, 30 minutes after the run, and 1-, 24-, 48, and 72-hours after the run.
  Interventions: Other: Running
- Cycling Group (Active Comparator): Participants cycle 39 kilometers. Venous blood is drawn prior to cycling, immediately after cycling, 30 minutes after cycling, and 1-, 24-, 48, and 72-hours after cycling.
  Interventions: Other: Cycling
- Rugby Group (Active Comparator): Participants play one rugby match. Venous blood is drawn prior to the match, immediately after the match, 30 minutes after the match and 1-, 24-, 48, and 72-hours after the match.
  Interventions: Other: Rugby
- Control Group (Placebo Comparator): Participants refrained from exercise for 24 hours followed by one blood draw.
  Interventions: Other: control group

INTERVENTIONS:
Other: Running — Participants were expected to run 6.44 kilometers.
  Other Names: Jogging
  Arms: Running Group
Other: Cycling — Participants were expected to cycle 39 kilometers
  Other Names: Biking
  Arms: Cycling Group
Other: Rugby — Participants were expected to play in one rugby match.
  Arms: Rugby Group
Other: control group — Participants were asked to refrain from exercise for 24 hours.
  Other Names: Control
  Arms: Control Group

SUMMARY:
The goal of this clinical trial was to determine if and how the biomarkers neurofilament light (NfL), brain lipid binding protein (BLBP), and amyloid precursor protein (APP) accumulated over 72 hours in venous blood following running, cycling, or playing rugby as compared to a non-exercising control group. Participants in this study were recreationally active and healthy males and females 18 - 49 years of age. The main questions it aimed to answer was:

Do NfL, BLBP, and APP increase following exercise? Researchers compared the accumulation of NfL, BLBP, and NfL among runners, cyclists, rugby players, controls, and between sexes in each category.

Participants were asked to either run, bike, play a rugby match, or abstain from exercise. In the exercising group, blood was drawn from a vein prior to the activity, immediately after the activity, 30 minutes after the activity, 1 hour after the activity, 24 hours after the activity, 48 hours after the activity, and 72 hours after the activity. In the non-exercising group blood was drawn from a vein one time.

DETAILED DESCRIPTION:
Participants were recruited for this study from fall 2021 - spring 2022. Participants recruited to play in a rugby match were current members of the university men's and women's club rugby team. Running participants consisted of members of the university's men's and women's running teams as well as recreational runners. Cycling participants consisted of members of the university's cycling club as well as recreational cyclists. Male rugby athletes played two 40-minute halves while female rugby athletes played two 20-minute halves. These are typical match times for men's and women's rugby. Runners were asked to run 6.44 kilometers at their own pace, and cyclists were asked to cycle 39 kilometers at their own pace. A control group comprised of both sedentary and recreationally active individuals was also recruited and asked to refrain from exercise for 24 hours.

Blood was drawn from an antecubital vein in the exercising groups before and after exercise as well as 30 minutes, 1-, 24-, 48-, and 72-hours after exercise. Only one blood draw was taken in the control group.

The blood biomarkers neurofilament light (NfL), brain lipid binding protein (BLBP), and amyloid precursor protein were then measured in the venous blood and compared within groups, among groups, and between sexes.

ELIGIBILITY:
Inclusion Criteria:

* Apparently Healthy
* Those in the running group must be able to run 6.44 kilometers
* Those in the cycling group must be able to cycle 39 kilometers
* Those in the ruby group must be members of the university club rugby team

Exclusion Criteria:

* Individuals with diabetes
* Individuals with heart disease
* Individuals who are pregnant
* Individuals who get light-headed or dizzy while donating blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Blood Biomarkers | Baseline, 0, 0.5, 1, 24, 48, 72 hours post-intervention.
  Neurofilament light (NfL) was measured in venous blood samples collected from participants. NfL was measured using enzyme-linked immunosorbent assays (ELISAs) in pg·mL-1.
Blood Biomarkers | Baseline, 0, 0.5, 1, 24, 48, 72 hours post-intervention.
  Brain lipid binding protein (BLBP) was measured in venous blood samples collected from participants. BLBP was measured using enzyme-linked immunosorbent assays (ELISAs) in ng·mL-1.
Blood Biomarkers | Baseline, 0, 0.5, 1, 24, 48, 72 hours post-intervention.
  Amyloid precursor protein (APP) was measured in venous blood samples collected from participants. APP was measured using enzyme-linked immunosorbent assays (ELISAs) in ng·mL-1.

CONTACTS AND LOCATIONS:
Locations (1):
- Appalachian State University, Boone, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The data set is small and collected from a specific population. Sharing IPD may indirectly identify some subjects.